CLINICAL TRIAL: NCT04423003
Title: Impact of the COVID-19 Pandemic on an Interdisciplinary Endoscopy Unit in a German "Hotspot" Area: a Single Center Experience
Brief Title: Endoscopic Interventions in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 242/2020BO2
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Change; Endoscopy, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic intervention — All endoscopic interventions in COVID-19 positive tested patients were included

SUMMARY:
This is a combined study including a descriptive part about the preparations for COVID-19 and the impact of COVID-19 on the daily routine of the work in an Interdisciplinary Endoscopic Unit (IEU), and a point-prevalence analysis for possible positive SARS-CoV-2 carriers among the staff of the IEU, and finally a prospective analysis of SARS-CoV-2 positive patients who required endoscopic intervention.

Results are presented in the captures: 1. SARS-CoV-2-pandemic related restructuring of the processes in the IEU, 2. SARS-CoV-2-pandemic related impact on the staff of the IEU, and 3. Analysis of endoscopic interventions in patients with confirmed or suspected SARS-CoV-2 infection.

DETAILED DESCRIPTION:
This article is intended to provide an overview of the impact of the COVID-19 pandemic on an interdisciplinary endoscopy unit (IEU, gastroenterological endoscopy, surgical endoscopy, and bronchoscopy) at the University Hospital Tübingen, a center for tertiary care in South-western Germany. First, preparations for COVID-19 pandemic with respect to the IEU are presented, and compared with those of other endoscopy units (7, 8). Additionally, the direct impact of SARS-CoV-2 on the staff of the IEU will be shown, together with a point-prevalence analysis of SARS-CoV-2 of the staff at the end of the SARS-CoV-2 wave in Tübingen. Finally, to our knowledge for the first time, we conducted a prospective single center analysis of the patients infected with SARS-CoV-2, which required a diagnostic or therapeutic endoscopic intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with proven or suspected infections with SARS-CoV-2 infection, who required endoscopic interventions

Exclusion Criteria:

* all other patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 10 patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
death in time of observation | 01.March 2020 to 5. May 2020
  death in time of observation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided